CLINICAL TRIAL: NCT02194621
Title: A Randomized, Single Center, Three Cell, Double Blind and Parallel Groups Clinical Study Conducted in Newark, NJ to Evaluate the Antibacterial Effects of Two Toothpastes Containing 0.3% Triclosan/2% Copolymer/0.243% Sodium Fluoride in a Silica Base as Compared to a Control Regular Fluoride Toothpaste on Oral Bacteria 12 Hours After 13 Days Product Use.
Brief Title: Clinical Investigation to Examine Toothpaste Effect on Oral Bacteria
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Colgate Palmolive (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CRO-1113-BACT-PS-NJ
Record Dates: First submitted 2014-07-15; First posted 2014-07-18 (Estimated); Results first posted 2016-04-15 (Estimated); Last update posted 2016-04-15 (Estimated); Status verified 2014-07

CONDITIONS: Oral Bacteria Levels in the Mouth
MeSH Terms: interventions — hydrated silica gel-based toothpaste

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Total Flavor Option 1 (Experimental): Total toothpaste containing triclosan/copolymer/sodium fluoride with new OM (oral malodor) complex 1 ingredient - Total Flavor Option 1
  Interventions: Drug: Total Flavor option 1
- Total Flavor Option 2 (Experimental): Total toothpaste containing triclosan/copolymer/sodium fluoride with new OM (oral malodor) complex 2 ingredient. Total Flavor Option 2
  Interventions: Drug: Total Flavor option 2
- Crest Toothpaste (Placebo Comparator): Placebo toothpaste: Crest Cavity Protection toothpaste (currently marketed)
  Interventions: Drug: Placebo toothpaste: Crest Cavity Protection toothpaste

INTERVENTIONS:
Drug: Total Flavor option 1 — Total toothpaste containing triclosan/copolymer/sodium fluoride with new OM complex 1 ingredient -Total Flavor Option 1
  Other Names: Total toothpaste
  Arms: Total Flavor Option 1
Drug: Total Flavor option 2 — Total toothpaste containing triclosan/copolymer/sodium fluoride and new OM complex 2 ingredient. Total Flavor option 2
  Other Names: Total toothpaste
  Arms: Total Flavor Option 2
Drug: Placebo toothpaste: Crest Cavity Protection toothpaste — Placebo toothpaste: Crest Cavity Protection toothpaste w/sodium fluoride (currently marketed)
  Other Names: Crest Anti-Cavity toothpaste
  Arms: Crest Toothpaste

SUMMARY:
The primary objective was to evaluate the antibacterial effects of two toothpastes containing 0.3% triclosan, 2% copolymer and 0.234% sodium fluoride in a silica base as compared to a control regular fluoride toothpaste on anaerobic and malodor bacteria 12 hours after 13 days of product use. A secondary objective was to demonstrate that a toothpaste containing 0.3% triclosan, 2% copolymer, 0.234% sodium fluoride and a flavor with odor-masking ingredients in silica base (Colgate Total Toothpaste-Flavor Option 1) provides a level of antibacterial efficacy that is "equivalent" to a toothpaste containing 0.3% triclosan, 2% copolymer, 0.234% sodium fluoride and a regular flavor in silica base (Colgate Total Toothpaste-Flavor Option 2) after 13 days of product use.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females in good general health aged 18 to 70 years.
2. A willingness to read, understand, and sign the Informed Consent Form after the nature of the study has been fully explained to them. Subject should demonstrate a willingness to comply with all study procedures and sampling schedules.
3. A minimum of 20 natural teeth with facial and lingual scorable surfaces.
4. Adequate oral hygiene and no signs of oral neglect.
5. Good periodontal health. Enrolled subjects will have no more than five periodontal pockets of 5 mm.
6. Subjects with gingival index greater than or equal to 1.0 (Loe-Silness Index) and plaque index greater than or equal to 1.5 (Turesky modification of Quigley-Hein Index) will be enrolled.

Exclusion Criteria:

1. History of significant adverse effects following use of oral hygiene products such as toothpastes and mouthrinses. Allergy to personal care/consumer products or their ingredients.
2. Teeth that are grossly carious, fully crowned or extensively restored on facial and/or lingual surfaces, orthodontically banded, abutments, or third molars
3. History of diabetes or hepatic or renal disease, or other serious medical conditions or transmittable diseases, e.g. heart disease or AIDS.
4. History of rheumatic fever, heart murmur, mitral valve prolapse or other conditions requiring prophylactic antibiotic coverage prior to invasive dental procedures.
5. Subjects on antibiotic, anti-inflammatory or anticoagulant therapy during the month preceding the baseline exam.
6. Significant oral soft tissue pathology, systemically related gingival enlargement, severe gingivitis (based on a visual examinations).
7. History of active severe periodontal disease with bleeding gums and loose teeth.
8. Gross dental caries, severe generalized cervical abrasion and/or enamel abrasion, large fractured or temporary restorations (based on visual examinations).will not be included in the tooth count.
9. Fixed or removable orthodontic appliance or removable partial dentures.
10. Participation in a dental plaque/gingivitis clinical study involving oral care products, within the last 30 days. History of dental prophylaxis or treatments in the past month.
11. Self reported pregnancy or lactation.
12. History or current use of objects to pierce the lips or tongue.
13. Subjects known to be an alcoholic, or a recovering alcoholic.
14. History or current use of recreational drugs.

Ages: 22 Years to 58 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 128 (Actual)
Dates: Start 2014-01; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Rutgers School of Dental Medicine, Newark, New Jersey, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: subject recruitment is completed locally at the clinical site
Pre-assignment Details: There will be a one (1) week wash out phase with commercially available fluoride toothpaste prior to any study intervention being assigned.
Groups:
- Total Flavor Option 1: Total toothpaste containing triclosan/copolymer/sodium fluoride with new OM complex 1 ingredient - Total Flavor Option 1
  Total Flavor option 1: Total toothpaste containing triclosan/copolymer/sodium fluoride with new OM complex 1 ingredient -Total Flavor Option 1
- Total Flavor Option 2: Total toothpaste containing triclosan/copolymer/sodium fluoride with new OM complex 2 ingredient. Total Flavor Option 2
  Total Flavor option 2: Total toothpaste containing triclosan/copolymer/sodium fluoride and new OM complex 2 ingredient. Total Flavor option 2
Period: Overall Study
Arm/Group | Total Flavor Option 1 | Total Flavor Option 2 | Crest Toothpaste
Started | 43 | 42 | 43
Completed | 37 | 36 | 34
Not Completed | 6 | 6 | 9
Not completed — 6 withdrew prior to randomization | 2 | 2 | 2
Not completed — Withdrawal by Subject | 4 | 4 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Total Flavor Option 1 | Total Flavor Option 2 | Crest Toothpaste | Total
Number analyzed (Participants) | 43 | 42 | 43 | 128
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.6 (10.2) | 34.2 (10.34) | 35.9 (12.08) | 35.4 (10.82)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 29 | 24 | 81
  Male | 15 | 13 | 19 | 47
Region of Enrollment [Number; unit: participants]
  United States | 43 | 42 | 43 | 128

OUTCOME MEASURES:

1. Primary Outcome: Anaerobic Bacteria
Description: Subjects brush their teeth with assigned toothpaste 2x/day for 13 days. On clinic visit day, subjects brush their teeth and return 12 hours later for clinical evaluation. Samples of dental plaque at the gumline will be collected for microbiological analysis to determine total levels of anaerobic bacteria CFU - colony forming units.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: colony forming units
Arm/Group | Total Flavor Option 1 | Total Flavor Option 2 | Crest Toothpaste
Number analyzed (Participants) | 43 | 42 | 43
colony forming units | 8.40 (0.33) | 8.42 (0.25) | 8.43 (0.28)
Statistical Analysis 1: Comparison: Total Flavor Option 1 vs Total Flavor Option 2 vs Crest Toothpaste; The null hypothesis states that there is no difference between groups; Test type: Superiority or Other; p > 0.05, ANOVA

2. Primary Outcome: Anaerobic Bacteria
Description: as for outcome 1
Time Frame: 12 hours
Measure: Mean (Standard Error); unit: colony forming units
Arm/Group | Total Flavor Option 1 | Total Flavor Option 2 | Crest Toothpaste
Number analyzed (Participants) | 37 | 36 | 34
colony forming units | 7.68 (0.09) | 7.71 (0.09) | 8.37 (0.09)
Statistical Analysis 1: Comparison: Total Flavor Option 2 vs Crest Toothpaste; The null hypothesis states that there is no difference between groups; Test type: Superiority or Other; p < 0.001, ANCOVA

3. Primary Outcome: Malodor Bacteria (Breath Odor Causing Bacteria)
Description: Subjects brush their teeth with assigned toothpaste 2x/day for 13 days. On clinic visit day, subjects brush their teeth and return 12 hours later for clinical evaluation. Samples of dental plaque at the gumline will be collected for microbiological analysis to determine levels of mouth odor causing bacteria CFU - colony forming units.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: colony forming units
Arm/Group | Total Flavor Option 1 | Total Flavor Option 2 | Crest Toothpaste
Number analyzed (Participants) | 37 | 36 | 34
colony forming units | 6.26 (0.44) | 6.26 (0.50) | 6.40 (0.46)
Statistical Analysis 1: Comparison: Total Flavor Option 1 vs Total Flavor Option 2 vs Crest Toothpaste; The null hypothesis states that there is no difference between groups; Test type: Superiority or Other; p > 0.05, ANOVA

4. Primary Outcome: Malodor Bacteria (Breath Odor Causing Bacteria)
Description: as for outcome 3
Time Frame: 12 hours
Measure: Mean (Standard Error); unit: colony forming units
Arm/Group | Total Flavor Option 1 | Total Flavor Option 2 | Crest Toothpaste
Number analyzed (Participants) | 37 | 36 | 34
colony forming units | 5.99 (0.07) | 5.92 (0.07) | 6.32 (0.07)
Statistical Analysis 1: Comparison: Total Flavor Option 1 vs Total Flavor Option 2 vs Crest Toothpaste; The null hypothesis states that there is no difference between groups; Test type: Superiority or Other; p = 0.002, ANCOVA

ADVERSE EVENTS:
Time Frame: Baseline, 12 hours and 2 weeks
Arm/Group | Total Flavor Option 1 | Total Flavor Option 2 | Crest Toothpaste
Serious Adverse Events (participants affected / at risk) | 0/43 | 0/42 | 0/43
Other Adverse Events (participants affected / at risk) | 0/43 | 0/42 | 0/43

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days